CLINICAL TRIAL: NCT06953297
Title: Exploring Vasopressin Use in Septic Shock: A Retrospective Cohort Study From Türkiye
Brief Title: Vasopressin Use in Septic Shock From Türkiye
Acronym: (VASCO-TURK)
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, A. Oguzhan KUCUK, Intensivist, Assistant Professor, Karadeniz Technical University
Other Study IDs: 2025-5
Record Dates: First submitted 2025-04-17; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Septic Shock; Vasodilatory Shock; Critical Illness Sepsis, Severe; Critical Illness; Intensive Care Medicine; Vasopressor Therapy
Keywords: Septic Shock; Vasopressin; Norepinephrine; Vasopressor Therapy; Hemodynamic Response; ICU; Critical Care; intensive care unit; Mortality; Lactate; Mean Arterial Pressure; Türkiye
MeSH Terms: conditions — Shock, Septic; Critical Illness; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Norepinephrine Only: Participants with septic shock who received norepinephrine as the sole vasopressor agent during their ICU stay. No adjunctive vasopressin or other vasopressors were administered. This group served as the reference for comparison of hemodynamic and clinical outcomes.
- Norepinephrine Plus Vasopressin: Participants with septic shock who received adjunctive vasopressin in addition to norepinephrine. Vasopressin was initiated during the course of vasodilatory shock based on clinical judgment. The study evaluated hemodynamic response and mortality in this group compared to norepinephrine monotherapy.

SUMMARY:
The goal of this observational study is to examine the early hemodynamic effects and clinical outcomes of vasopressin use in patients with septic shock. The study aims to compare adult ICU patients who received norepinephrine alone versus those who received vasopressin in addition to norepinephrine.

The main question it aims to answer is:

Does adding vasopressin to norepinephrine improve blood pressure, lactate levels, and survival in patients with septic shock?

Researchers used retrospective medical records of patients treated between January and December 2024. Data such as blood pressure, heart rate, lactate levels, and mortality were collected and analyzed to assess treatment response and outcomes.

DETAILED DESCRIPTION:
This is a single-center, retrospective observational cohort study designed to evaluate the clinical impact of adjunctive vasopressin therapy in adult patients with septic shock. The study protocol was developed to assess early hemodynamic responses and mortality outcomes associated with vasopressin use in real-world intensive care settings in Türkiye.

A total of 146 adult patients admitted to the intensive care unit (ICU) between January 1 and December 15, 2024, were included in the study. All patients fulfilled Sepsis-3 criteria for septic shock and received norepinephrine as the primary vasopressor agent. Among these, 33 patients received vasopressin in addition to norepinephrine, while the remaining patients were managed with norepinephrine alone.

The primary objective of the study is to describe early hemodynamic changes following vasopressin administration, specifically focusing on changes in:

Mean arterial pressure (MAP),

Heart rate (HR),

Serum lactate levels, and

Norepinephrine dose requirement,

within the first 6 and 24 hours of vasopressin initiation.

The secondary objective is to assess all-cause mortality among patients who received norepinephrine alone versus those treated with norepinephrine plus vasopressin.

All data were collected retrospectively from the institution's electronic health record system. Patients who received dopamine or epinephrine either prior to or concurrently with vasopressin were excluded to ensure homogeneity of the treatment groups. No randomization or prospective allocation was involved, and all treatment decisions were made by the clinical ICU team as part of routine medical care.

Statistical analyses will include descriptive and inferential methods to compare outcomes between the two groups, including Mann-Whitney U test, Chi-square test, Friedman's test, and Kaplan-Meier survival analysis. This study aims to describe the protocol and methodology of a real-world, retrospective analysis and does not intend to present prospective results at this stage.

The protocol was approved by the institutional ethics committee and adheres to international standards for human subject research.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) admitted to the intensive care unit (ICU)
* Diagnosed with septic shock according to Sepsis-3 criteria
* Treated with norepinephrine as the initial vasopressor
* Received norepinephrine alone or norepinephrine with adjunctive vasopressin
* Admitted between January 1 and December 15, 2024

Exclusion Criteria:

* Patients younger than 18 years
* Patients who received epinephrine or dopamine prior to or along with vasopressin
* Patients with incomplete clinical or hemodynamic data
* Readmitted ICU patients during the same hospitalization
* Patients with do-not-resuscitate (DNR) orders at ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients with septic shock admitted to the intensive care unit of a tertiary academic hospital in Türkiye. All participants received norepinephrine as a first-line vasopressor, and a subset received adjunctive vasopressin.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Mean Arterial Pressure (MAP) Within 24 Hours After Vasopressin Initiation | 6 hours after vasopressor initiation
  Mean arterial pressure (MAP) will be recorded at vasopressin initiation and at 0, 2 and 6 hours following the first dose. The primary outcome is the absolute change in MAP from baseline to 24 hours in patients receiving adjunctive vasopressin compared to those receiving norepinephrine alone.

SECONDARY OUTCOMES:
All-Cause Mortality | Up to Day 28 after ICU admission
  Vital status (alive or deceased) at day 28 after ICU admission will be collected from medical records to compare mortality between treatment groups.
Change in Serum Lactate Levels | 6 hours
  Serum lactate concentrations will be measured at vasopressin initiation, and at 0, 2 and 6 hours. The study will assess reductions in lactate as a marker of improved perfusion.
Change in Norepinephrine Dose After Vasopressin Initiation | 6 hours
  Norepinephrine infusion dose (mcg/kg/min) will be measured at vasopressin initiation and at 0, 2 and 6 hours. The outcome is the reduction in dose over time indicating vasopressor-sparing effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Faculty of Medicine, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The dataset includes identifiable patient-level clinical data from a retrospective ICU cohort. Due to ethical and privacy considerations, individual participant data (IPD) will not be shared.

REFERENCES:
- [Derived] Kucuk AO, Hocek AB, Aydin D, Acar B, Pehlivanlar E, Pehlivanlar Kucuk M. Exploring vasopressin use in septic shock: a retrospective cohort study from Turkiye (VASCO-TURK). BMC Anesthesiol. 2025 Nov 22;25(1):623. doi: 10.1186/s12871-025-03519-8. PMID 41275079